CLINICAL TRIAL: NCT00535067
Title: Neuropathic Pain in Survivors of Breast Cancer
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 2006-0761
Record Dates: First submitted 2007-09-21; First posted 2007-09-26 (Estimated); Last update posted 2015-01-09 (Estimated); Status verified 2015-01

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Questionnaire; Survey; Neuropathic Pain; Cancer Survivors; Quality of Life; QOL
MeSH Terms: conditions — Breast Neoplasms; Neuralgia | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Breast Cancer Survivors
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Questionnaires taking 60 minutes total to complete.
  Other Names: Survey

SUMMARY:
The objectives of this study are to: 1) describe the prevalence of neuropathic pain (NP) in breast cancer survivors and 2) to develop preliminary statistical risk models for predicting the risk for NP incorporating disease-related variables (e.g., stage of disease, location of tumor), treatment variables (chemotherapy, dose, duration; and other cancer therapy), clinical health status (e.g., comorbid conditions), and sociodemographic characteristics (e.g., age, sex, race).

Researchers will also gather data to answer the following secondary aims:

1. To assess the impact of NP on quality of life.
2. To assess the current management of NP in cancer (current medication, duration of such treatment, reasons for discontinuation) and the outcomes of this management.

DETAILED DESCRIPTION:
You have already been contacted by phone about participating in this study. You have received study documents (this consent and the study questionnaires) because you said over the phone that you would like to participate in this study.

In this study you will be asked to complete questionnaires that will ask about any pain you may be experiencing and about the quality of your life. These questionnaires will also ask for demographic information (such as age, race, and sex) and about your health. It should take about 1 hour to complete all of the questionnaires. In addition to the questionnaires, you will also be asked questions about any medications you may currently be taking for pain. All of the information you include on the questionnaires will be kept confidential. There are no right or wrong answers to the questions. A postage-paid return envelope has been provided for you to return this consent and the questionnaires.

Researchers are interested in how pain is related to certain treatments and medical conditions. As part of this study, researchers will review your medical records to see what type of cancer treatment you received and whether you had any pain related to the treatment. They will also see if you had any non-cancer health conditions that may have affected pain and quality of life.

This survey is for research purposes only. Your healthcare provider will not be informed of your responses to this survey. If you are experiencing severe pain and/or other symptoms, please contact your healthcare provider. The study staff has also included a list of community resources that you may contact for different types of services.

Your participation in this study will be over once you mail back the consent and questionnaires.

This is an investigational study. Up to 635 individuals will be asked to take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients who were participants in clinical trials (ID98-240; ID94-002) for taxanes during 1994-2001
* Alive and with current contact information
* Age ≥ 18 years. (This restriction is based on inclusion criteria for the clinical trials from which subjects will be recruited. All patients will be at least 18 years or older for this study.)

Exclusion Criteria:

1) None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast Cancer survivors.
Sampling Method: Non-Probability Sample
Enrollment: 239 (Actual)
Dates: Start 2007-09; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Prevalence of neuropathic pain (NP) in breast cancer survivors | 3 Years
  Assessment of neuropathic pain will be standardized using two validated tools for this purpose: the self report version of the LANSS pain score (S-LANSS) [Bennett 2001, Bennett et al 2004] and ID Pain (IDP) [Portenoy, et al, 2006]. The S-LANSS is a 7-item instrument that identifies pain of predominantly neuropathic origin. A score of 10 or more (out of a maximum of 24), regarded as a "positive" score, identifies neuropathic pain with a sensitivity, specificity and positive predictive value all of 80%. It has been found to be valid and reliable in both clinical and mail-survey settings [Bennett et al 2004]. The IDP is a 6-item scale that assesses the quality of pain, and has been well-validated [Portenoy, et al, 2006].

SECONDARY OUTCOMES:
Study of how much pain, factors related to the pain, and how the pain affects life | 3 Years
  Preliminary statistical risk models for predicting the risk for NP incorporating disease-related variables (e.g., stage of disease, location of tumor), treatment variables (chemotherapy, dose, duration; and other cancer therapy), clinical health status (e.g., comorbid conditions), and sociodemographic characteristics (e.g., age, sex, race).

CONTACTS AND LOCATIONS:
Overall Officials: Cielito C. Reyes-Gibby, DrPH, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org